CLINICAL TRIAL: NCT04344327
Title: Early Risk Stratification of Patient Hospitalized for SARS-CoV2 Infection: Critical COVID-19 France CCF
Acronym: CCF
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020-02
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Infection Viral; Infection, Hospital; COVID
Keywords: Cardiology department; Medicine conventional department
MeSH Terms: conditions — Virus Diseases; Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with COVID-19: Patients hospitalized in conventional sector with diagnosis of COVID-19 (positive PCR (Polymerase Chain Reaction) or diagnosis presumed by the clinical and radiographic picture)

SUMMARY:
The COVID-19 pandemic of SARS CoV2 (Severe Acute Respiratory Syndrome, COVID-19) infection, which is currently evolving in France, raises many questions about the clinical and biological profile of infected hospitalized patients. If certain biological factors like troponin, BNP (Brain Natriuretic Peptid), or clinical factors like cardiovascular history or oncological history are associated with a worse prognosis, available data comes from studies in Asia for the majority, or including a limited number of patients. Patient stratification remains a major issue for patient sorting and early referral of patients.

DETAILED DESCRIPTION:
This study is observational, multicenter and retrospective, and is conducted in hospitals in France.

Clinical data relating to history, comorbidities, risk factors, previous treatments, treatments during the hospitalization and treatments at the discharge from hospital, clinical parameters, biological and ultrasound cardiological data, procedures and events during hospitalization will be recorded, in order to identify the early predictors of clinical worsening in patients hospitalized for COVID-19 in cardiology or conventional medicine department.

ELIGIBILITY:
Inclusion Criteria:

- Patients hospitalized in cardiology unit or medicine conventional sector with diagnosis of COVID-19 (positive PCR (Polymerase Chain Reaction) or diagnosis presumed by the clinical and radiographic picture)

Exclusion Criteria:

* Minors
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the hospital with COVID-19 infection
Sampling Method: Probability Sample
Enrollment: 2878 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Death rate | Through study completion, an average of 4 weeks
  Analysis of all-cause death in relation with clinical patient profile
Transfer to intensive care unit | Through study completion, an average of 4 weeks
  Correlation between clinical patient profile and transfer need to intensive care unit
Ventilation analysis | Through study completion, an average of 4 weeks
  Type of ventilation procedures needed during the hospitalization (Orotracheal intubation for mechanical ventilation or Non-invasive ventilation or 29/5000 high flow oxygen therapy - Optiflow) in relation with clinical patient profile

SECONDARY OUTCOMES:
Construction of a predictive score for COVID-19 severe form | Through study completion, an average of 4 weeks
  Description of clinical and biological patient profile leading to a worse prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume BONNET, MD, Study Director — Hopital Européen Georges Pompidou; Orianne WEIZMAN, MD, Principal Investigator — Central Hospital, Nancy, France
Locations (23):
- France (23):
  - CHU d'Amiens, Amiens
  - CHU Annecy, Annecy
  - CHU de Bordeaux, Bordeaux
  - CHU de Caen, Caen
  - Cotentin hospital, Cherbourg
  - CHU Dijon, Dijon
  - Elbeuf Louviers Val de Reuil, Elbeuf
  - CHU de Fréjus / Saint-Raphael, Fréjus
  - Lille Catholic Institute Hospital Group, Lille, Lille
  - CHU de Lyon, Lyon
  - APHM, Marseille
  - Jacques Cartier Private Hospital, Massy, Massy
  - CHR d'Orléans, Orléans
  - Bichat (APHP), Paris
  - Georges Pompidou European Hospital (AP-HP), Paris
  - Institut Mutualiste Montsouris, Paris, Paris
  - CHU de Reims, Reims
  - CHU de Rouen, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - Saint Gatien hospital, Tours
  - CHU de Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sutter W, Duceau B, Vignac M, Bonnet G, Carlier A, Roussel R, Trimaille A, Pommier T, Guilleminot P, Sagnard A, Pastier J, Weizman O, Giordano G, Cellier J, Geneste L, Panagides V, Marsou W, Deney A, Karsenty C, Attou S, Delmotte T, Ribeyrolles S, Chemaly P, Gautier A, Fauvel C, Chaumont C, Mika D, Pezel T, Cohen A, Potier L; Critical COVID-19 France Investigators. Association of diabetes and outcomes in patients with COVID-19: Propensity score-matched analyses from a French retrospective cohort. Diabetes Metab. 2021 Jul;47(4):101222. doi: 10.1016/j.diabet.2020.101222. Epub 2020 Dec 31. PMID 33388386